CLINICAL TRIAL: NCT01246297
Title: A Pilot Study of Early Outpatient Pulmonary Rehabilitation Following Thoracic Surgery for Lung Cancer
Brief Title: Effect of Pulmonary Rehabilitation in Lung Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College Healthcare NHS Trust (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other); London Cancer Alliance (North West London Cancer Network) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JROSM0090
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Lung Cancer; Lobectomy; Pulmonary Rehabilitation
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Other): Usual Care
  Interventions: Other: Usual post operative care
- Pulmonary Rehabilitation (Active Comparator): Pulmonary Rehabilitation consists of twice weekly exercise classes with an educational component.
  Interventions: Other: Pulmonary Rehabilitation

INTERVENTIONS:
Other: Pulmonary Rehabilitation — Twice weekly exercise classes with an education component. For 8 weeks.
  Arms: Pulmonary Rehabilitation
Other: Usual post operative care — Usual post operative care for post lung lobectomy patients for 8 weeks post discharge.
  Arms: Control

SUMMARY:
Patients who have surgery to cure lung cancer often have multiple problems at hospital discharge and later on. This includes poor exercise performance and quality of life, breathlessness, pain and tiredness. Currently there is little formal physical or psychological support for such patients. This pilot study aims to investigate whether outpatient pulmonary rehabilitation (an exercise training and education programme), started within 2 weeks of hospital discharge, can lead to improvements in exercise performance and quality of life in patients who have undergone lung cancer surgery. The study will also assess whether pulmonary rehabilitation is acceptable for patients and will analyze the safety profile. The hypothesis is that patients; discharged from hospital after undergoing lung cancer surgery, have improved exercise performance and quality of life following early outpatient pulmonary rehabilitation compared with usual care.

DETAILED DESCRIPTION:
The research question is to investigate

* whether patients who have undergone curative surgical resection for lung cancer benefit from 8 weeks of early outpatient pulmonary rehabilitation (started within 2 weeks of hospital discharge).
* to identify potential barriers to this approach

Pulmonary rehabilitation (PR) is the most effective non-pharmacological treatment for patients with chronic respiratory diseases, especially COPD. Many patients with lung cancer have co-existing smoking-related lung disorders such as COPD. To date there have been no randomised controlled trials of PR in post-resection lung cancer survivors. However there is indirect evidence that PR may be of benefit in this patient cohort. Cesario et al (2007)reported a 32% improvement in exercise capacity with in-patient PR, and Spruit et al (2009) demonstrated a 43% improvement in six minute walk distance following an 8-week in-patient PR programme. However, both studies had small numbers, and no randomised control group. Furthermore, inpatient PR is not an economically justifiable intervention in the NHS where emphasis is on self-management and ambulatory care.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing lung cancer surgery with curative intent.

Exclusion Criteria:

* Unstable cardiovascular disease Severe musculo-skeletal problems that would limit exercise training(neuromuscular disorders, severe joint arthritis of lower limbs) Severe peripheral vascular disease Unable to walk 10 metres unaided Patients unable to give informed consent Recent (within 3 months of completing treatment) or untreated pulmonary TB, Untreated/uncontrolled diabetes or epilepsy Recent or recurrent untreated spontaneous pneumothorax

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-10; Primary Completion 2011-07 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Six minute walk test to assess exercise tolerance | Within 3 month of discharge from surgery

SECONDARY OUTCOMES:
Shoulder Range of Motion Changes | Within 3 months of discharge from surgery
Bioimpedence for tissue composition | Within 3 months of discharge from surgery
Quality of life measurement changes | Within 3 months of discharge from surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Elkin, FRCP, Principal Investigator — Imperial College Healthcare Trust
Locations (2):
- United Kingdom (2):
  - Harefield Hospital, Harefield, Middlesex
  - Imperial College Healthcare Trust, London